CLINICAL TRIAL: NCT01847170
Title: Impact of Fecal Biotherapy (FBT) on Microbial Diversity in Patients With Moderate to Severe Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: The Broad Foundation (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Alan C. Moss, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P000353
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbial Transplantation (Experimental)
  Interventions: Biological: Fecal Microbial Transplantation

INTERVENTIONS:
Biological: Fecal Microbial Transplantation
  Other Names: Fecal Transplant; Stool transplant

SUMMARY:
The human immune system is usually tolerant of the millions of beneficial commensal bacteria (the microbiome), which colonize the healthy intestinal tract. In contrast, patients with Inflammatory Bowel Disease (IBD) may play host to an imbalanced mix of such intestinal bacteria, which initiates abnormal immune responses in susceptible individuals. The resulting inflammation that occurs in the gastrointestinal tract damages the intestinal lining, leading to symptoms (such as intractable diarrhea, pain or weight loss), heightened cancer risk, other serious complications with substantial morbidity and even death. Current therapies for IBD focus on suppressing the excessive immune response to these bacteria, but have major side effects and do not address any role of the microbiome in disease development.

The investigators hypothesize that there is heightened intraluminal generation of pro-inflammatory factors by luminal "pathogenic" bacteria, such as extracellular nucleotides and purinergic derivatives, which trigger host immune cells. This results in loss of suppressive T regulatory cells with unrestrained immune cell deviation to pathogenic T helper cells that cause inflammatory responses. The investigators' proposal is that correcting the disease-provoking microbiome would beneficially improve gut microbial diversity, alter immune responses elicited in patients by such microbial products of pathogenic bacteria, and ultimately limit and suppress disease activity.

To test the hypothesis, the investigators propose to enroll patients with active Crohn's Disease, and introduce the microbiome of healthy and unrelated individuals to patient's intestinal tract, via fecal biotherapy (FBT) with all applicable safety measures. The investigators propose to comprehensively test the effects of FBT on the host microbiome, determine microbial production of inflammatory nucleotides and derivatives, which the investigators suggest might impact the host immune response and disease activity in patients with IBD.

ELIGIBILITY:
Inclusion Criteria (Patients):

* CD confirmed by biopsy for > 3 months duration
* Active disease (Harvey-Bradshaw Index > 5
* Failed standard therapy with; stable doses of 5-ASA >2 weeks; thiopurines >3 months; or is steroid dependent at a dose <20mg/d; (inability to taper off steroid for longer than 1 week)
* Stable medication regimen for >2 weeks.
* Age > 18 years old

Exclusion Criteria (Patients):

* Diagnosis of indeterminate colitis, or proctitis alone
* Severe or fulminate colitis
* Women who are pregnant or nursing
* Patients who are unable to give informed consent
* Patients who are unable or unwilling to undergo colonoscopy with moderate sedation (>ASA class II)
* Patients who have previously undergone FMT
* Patients who have a confirmed malignancy or cancer
* Patients who are immunocompromised
* Treatment within last 12 weeks with cyclosporine, tacrolimus, infliximab, adalimumab, certolizumab, natalizumab, thalidomide
* Antibiotic use within 2-months of start date
* Participation in a clinical trial in the preceding 30 days or simultaneously during this trial
* Probiotic use within 30 days of start date
* Rectal therapy within 14 days of start date
* Decompensated cirrhosis
* Congenital or acquired immunodeficiencies
* Other comorbidities including:
* Diabetes mellitus, cancer, systemic lupus, must be able to tolerate conscious sedation with colonoscopy
* Chronic kidney disease as defined by a GFR <60mL/min/1.73m2 44
* History of rheumatic heart disease, endocarditis, or valvular disease due to risk of bacteremia from colonoscopy
* Steroid dose >20mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety of FMT in patients with Crohn's disease, as measured by number and nature of adverse events | 24 weeks
Recipients' fecal microbial diversity after FMT, when compared to baseline | 12 weeks

SECONDARY OUTCOMES:
Recipients' fecal microbial diversity at 4 and 8 weeks after FMT, when compared to baseline | 8 weeks
Mean change in Harvey Bradshaw Index (HBI) score | 12 weeks
Percentage of patients in clinical remission (those with an HBI score at week 12 <5) | 12 weeks
Mean change in Short Inflammatory Bowel Disease Questionnaire (sIBDQ) score | 12 weeks
Percentage of patients in endoscopic remission (CDEIS score <3) | 12 weeks
Percentage of patients with mucosal healing (CDEIS score <1) | 12 weeks
Mean change in CRP levels | 12 weeks
Mean change in Crohn's Disease Endoscopic Index of Severity (CDEIS) score | 12 weeks
Tolerability score | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Moss, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Vaughn BP, Vatanen T, Allegretti JR, Bai A, Xavier RJ, Korzenik J, Gevers D, Ting A, Robson SC, Moss AC. Increased Intestinal Microbial Diversity Following Fecal Microbiota Transplant for Active Crohn's Disease. Inflamm Bowel Dis. 2016 Sep;22(9):2182-90. doi: 10.1097/MIB.0000000000000893. PMID 27542133